CLINICAL TRIAL: NCT00075998
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of the Safety and Efficacy of Interferon Gamma-1b in Patients With Idiopathic Pulmonary Fibrosis (The INSPIRE Trial)
Brief Title: The INSPIRE Trial: A Study of Interferon Gamma-1b for Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: test drug showed lack of benefit at interim analysis
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIPF-007
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Idiopathic Pulmonary Fibrosis; Lung Disease; Pulmonary Fibrosis
Keywords: Idiopathic; Pulmonary; Fibrosis; IPF; Lung; Interferon; Gamma; Actimmune; INSPIRE; InterMune
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases; Pulmonary Fibrosis; Fibrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interferon gamma-1b ("Actimmune") — 200 mcg, SQ, 3x per week

SUMMARY:
* Purpose: A phase 3, randomized, double-blind, placebo-controlled trial to determine the efficacy and safety of 200 µg of recombinant Interferon gamma-1b administered by subcutaneous (SC) injection, compared with placebo, in patients with IPF
* Enrollment: Approximately 800 patients will be enrolled from approximately 80 centers in North America and Europe
* Randomization: 2:1 active-to-placebo ratio
* Duration: at least 2 years active drug or placebo (rescue therapy will be permitted for patients who meet predefined criteria)

DETAILED DESCRIPTION:
INSPIRE, the largest and most comprehensive clinical trial ever conducted in IPF, has now completed enrolling patients with mild to moderate IPF. Eligible patients will receive either Interferon gamma-1b or placebo for a minimum of 2 years.

ELIGIBILITY:
Inclusion criteria:

* Clinical symptoms consistent with IPF of >= 3 months duration
* Diagnosis of IPF within 48 months before randomization
* Age 40 through 79, inclusive
* High-resolution computed tomographic scan (HRCT) showing definite IPF. For patients with surgical lung biopsy showing definite or probable usual interstitial pneumonia (UIP), the HRCT criterion of probable IPF is sufficient.
* For patients aged < 50 years: open or video-assisted thoracoscopic (VATS) lung biopsy showing definite or probable UIP within 48 months before randomization. In addition, there are no features supporting an alternative diagnosis on transbronchial biopsy or bronchoalveolar lavage (BAL) if performed.
* For patients aged < 50 years: At least one of the following diagnostic findings, as well as the absence of any features on specimens resulting from any of these procedures that support an alternative diagnosis, within 48 months before randomization:

  * Open or VATS lung biopsy showing definite or probable UIP
  * Transbronchial biopsy showing no features to support an alternative diagnosis
  * BAL showing no features to support an alternative diagnosis IPF Disease Severity and Progression
* FVC >= 55% of predicted value (post administration of bronchodilator)
* Hemoglobin (Hb)-corrected carbon monoxide diffusing capacity/carbon monoxide transfer capacity (DLCO/TLCO) >= 35% of predicted value
* At least one of either FVC or Hb-corrected DLCO/TLCO <= 90% of predicted value
* IPF disease progression evidenced by one or more of the following within the past year and the absence of evidence of improvement in the past year:

  * Absolute decrease of >= 10% in FVC
  * Absolute decrease of >= 15% in DLCO/TLCO
  * Evidence of clinically significant worsening on chest X ray or HRCT
  * Significant worsening of dyspnea
* Distance walked >= 150 meters (492 feet) with O2 saturation >= 83% on <= 6 L/min of O2 during the 6 Minute Walk Test (6MWT) oxygen titration procedure

Exclusion criteria:

1. Not a suitable candidate for enrollment or unlikely to comply with the requirements of this study, in the opinion of the Principal Investigator (PI)
2. Forced expiratory volume in the first second (FEV1)/FVC ratio < 0.6 (after administration of bronchodilator)
3. Residual volume (RV) > 140% of predicted (before administration of bronchodilator)
4. History of clinically significant environmental exposure known to cause pulmonary fibrosis (including but not limited to drugs, asbestos, beryllium, radiation, domestic birds)
5. Known explanation for interstitial lung disease, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, and cancer
6. Diagnosis of any connective tissue disease, including but not limited to scleroderma, systemic lupus erythematosus, and rheumatoid arthritis
7. Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, and cellulitis
8. On a lung transplantation waiting list at time of randomization

   Medical Exclusions:
9. Any history of malignancy likely to result in death, significant disability, or likely to require significant medical or surgical intervention within the next 3 years. This does not include minor surgical procedures for localized carcinoma (e.g., basal cell carcinoma)
10. Any condition other than IPF which, in the opinion of the PI, is likely to result in the death of the patient within the next 3 years
11. History of unstable or deteriorating cardiac, vascular, or neurologic disease within the previous 6 months, including but not limited to the following:

    * Myocardial infarction, unstable angina pectoris, coronary artery bypass surgery, or coronary angioplasty
    * Congestive heart failure requiring hospitalization
    * Uncontrolled arrhythmias
    * Thromboembolic event (e.g., deep vein thrombosis, pulmonary embolism)
    * Transient ischemic attacks (TIAs) or cerebral vascular accident
12. Any condition, which, in the opinion of the investigator, might be significantly exacerbated by the known side effects, (e.g., flu-like syndrome) associated with the administration of IFN g 1b
13. History of any of the following medical conditions:

    * Multiple sclerosis
    * Seizures within the past 10 years or taking anti seizure medication
    * Severe or poorly controlled diabetes
14. Pregnancy or lactation. Females of childbearing potential are required to have a negative serum pregnancy test before treatment and must agree to practice abstinence or prevent pregnancy by at least a barrier method of birth control for the duration of the study
15. Inability to tolerate nonsteroidal anti-inflammatory drugs (NSAIDS) or acetaminophen (paracetamol)
16. History of ethanol abuse in the past 2 years
17. Known hypersensitivity to IFN-g or closely related interferons or to any component of the study treatment
18. Presence of human immunodeficiency virus (HIV) or chronic viral hepatitis

    Laboratory Exclusions:
19. Any of the following liver function test criteria above specified limits:

    Total bilirubin > 1.5 x upper limit of normal (ULN); aspartate or alanine aminotransferases (AST/SGOT or ALT/SGPT) > 2 x ULN; alkaline phosphatase > 2 x ULN; or albumin < 3.0 mg/dL
20. Any of the following hematology test criteria outside of specified limits: WBC < 2,500/mm3, hematocrit < 30% or > 59%, platelets < 100,000 /mm3
21. Creatinine > 1.5 x ULN

    Concomitant Therapy Exclusions:
22. Prednisone therapy (prednisone or equivalent, with dose adjusted for potency) in excess of 0.125 mg/kg ideal body weight (IBW) per day or in excess of 0.25 mg/kg IBW every other day. Patients will also be excluded if they were not on a stable dose of corticosteroid therapy for at least 28 days prior to screening.
23. Prior treatment with IFN g 1b
24. Investigational therapy (i.e., agents that are not approved by local regulatory agencies) for any indication within 28 days prior to screening
25. The following therapies are excluded within 28 days prior to screening:

    * Investigational therapy for IPF, including pirfenidone
    * Any cytotoxic/immunosuppressive agent other than corticosteroids (including but not limited to azathioprine, cyclophosphamide, methotrexate, cyclosporine)
    * Any cytokine modulators (including but not limited to etanercept, infliximab)
    * Any therapy targeted to treat IPF (including but not limited to d penicillamine, colchicine, bosentan, N-acetyl-cysteine [NAC])

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2003-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Survival time from randomization to treatment completion visit, or, end of treatment period, or, last known vital status. | 3.5 years

SECONDARY OUTCOMES:
Lung transplant-free survival time (ongoing assessment up to end of study). | 3.5 years
Total number of days without hospitalization resulting from respiratory admission diagnosis (ongoing assessment up to end of study). | 3.5 years
Changes from baseline measurement to week 96 measurement in the following (measured every 24 weeks): 6-minute walk test, shortness of breath | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: InterMune, Inc., Study Chair — Medical Information
Locations (1):
- InterMune, Inc., Brisbane, California, United States

REFERENCES:
- [Derived] Wells AU, Jacob J, Sverzellati N, Cross G, Barnett J, De Lauretis A, Antoniou K, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. A formula for predicting emphysema extent in combined idiopathic pulmonary fibrosis and emphysema. Respir Res. 2024 Jan 18;25(1):33. doi: 10.1186/s12931-023-02589-x. PMID 38238788
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Kreuter M, Lee JS, Tzouvelekis A, Oldham JM, Molyneaux PL, Weycker D, Atwood M, Kirchgaessler KU, Maher TM. Monocyte Count as a Prognostic Biomarker in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2021 Jul 1;204(1):74-81. doi: 10.1164/rccm.202003-0669OC. PMID 33434107
- [Derived] Kreuter M, Lederer DJ, Molina-Molina M, Noth I, Valenzuela C, Frankenstein L, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. Association of Angiotensin Modulators With the Course of Idiopathic Pulmonary Fibrosis. Chest. 2019 Oct;156(4):706-714. doi: 10.1016/j.chest.2019.04.015. Epub 2019 Apr 29. PMID 31047956
- [Derived] Cottin V, Hansell DM, Sverzellati N, Weycker D, Antoniou KM, Atwood M, Oster G, Kirchgaessler KU, Collard HR, Wells AU. Effect of Emphysema Extent on Serial Lung Function in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1162-1171. doi: 10.1164/rccm.201612-2492OC. PMID 28657784
- [Derived] du Bois RM, Albera C, Bradford WZ, Costabel U, Leff JA, Noble PW, Sahn SA, Valeyre D, Weycker D, King TE Jr. 6-Minute walk distance is an independent predictor of mortality in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2014 May;43(5):1421-9. doi: 10.1183/09031936.00131813. Epub 2013 Dec 5. PMID 24311766
- [Derived] King TE Jr, Albera C, Bradford WZ, Costabel U, Hormel P, Lancaster L, Noble PW, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, du Bois RM; INSPIRE Study Group. Effect of interferon gamma-1b on survival in patients with idiopathic pulmonary fibrosis (INSPIRE): a multicentre, randomised, placebo-controlled trial. Lancet. 2009 Jul 18;374(9685):222-8. doi: 10.1016/S0140-6736(09)60551-1. Epub 2009 Jun 29. PMID 19570573